CLINICAL TRIAL: NCT03965416
Title: Influence of White Coat on Communication During General and Family Medicine Consultation: Interventional Study
Brief Title: Influence of White Coat During Family Medicine Consultation: Interventional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Leonor Marques Caetano Carreira, Student, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018.02
Record Dates: First submitted 2019-05-22; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Communication
Keywords: White Coat; Communication; Physician - Patient Relationship; Satisfaction; Trust; Competence; Empathy; Knowledge
MeSH Terms: conditions — Communication; Personal Satisfaction | interventions — White Coat tooth coating material

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doctor with white coat (Experimental): Doctor during consultation is wearing a white coat
  Interventions: Other: White Coat
- Doctor without white coat (Experimental): Doctor during consultation is not wearing a white coat
  Interventions: Other: Without White Coat

INTERVENTIONS:
Other: White Coat — We included the first and last patients in consultation every day for 10 consecutive days, and every other day the doctor consulted with the use of a white coat or without the use of a white coat.
  Arms: Doctor with white coat
Other: Without White Coat — We included the first and last patients in consultation every day for 10 consecutive days, and every other day the doctor consulted with the use of a white coat or without the use of a white coat.
  Arms: Doctor without white coat

SUMMARY:
Introduction: The white coat is a physician attire worn since the antiquity time. Several studies in other countries have shown that it influences doctor-patient's relationship and that there is some kind of preference over what a doctor should wear. In Portugal there are few data on this subject.

Objectives: Investigate the influence of the white coat on satisfaction, confidence and empathy in relation to patients. Secondly, its impact on what patients perceive about medical knowledge, patients' opinions about medical clothing, and the level of satisfaction and comfort of physicians in consultation with or without the use of a white coat.

Methods: An interventional study with a quasi-randomized representative sample of the population attending the health centers belonging to ARS Centro, consisting of 286 participants. The investigators collaborated with 16 doctors, male and female and of different ages which usually wore white coat in their medical appointments. The investigators included the first and last patients in consultation every day for 10 consecutive days, and every other day the doctor consulted with the use of a white coat or without the use of a white coat. At the end of the consultation, a questionnaire was distributed to the patient. This questionnaire had simple questions with a Lickert scale response, the portuguese version of the scale "Trust in physician" to assess the trust in the physician, both globally and in the medical-patient's relationship and their medical competences, and the JSPPPE-VP scale to evaluate empathy. A questionnaire was also distributed to the physician in which the doctor indicated what type of attire that used on that appointment and how satisfied and comfortable was with the consultation.

DETAILED DESCRIPTION:
1. INTRODUCTION

   The white coat is a physician attire worn since the antiquity time. Several studies in other countries have shown that it influences doctor-patient's relationship and that there is some kind of preference over what a doctor should wear. In Portugal there are few data on this subject.

   Objectives: Investigate the influence of the white coat on satisfaction, confidence and empathy in relation to patients. Secondly, its impact on what patients perceive about medical knowledge, patients' opinions about medical clothing, and the level of satisfaction and comfort of physicians in consultation with or without the use of a white coat.
2. METHODOLOGY

2.1 - Research characterization

An intervention study has been conducted evaluating the use or not of the white coat, in a quasi-random sample in the patient population attending health care centres in the central region of Portugal.

2.2 - Population, sample and exclusion criteria

The questionnaire was applied to a population sample calculated to represent, with a confidence interval of 90% and a margin of error of 5%, the population attending the consultations using the formula accessible at www.raosoft.com/samplesize.html (271 patients).

About 16 volunteer physicians were invited by the researchers to collaborate. These included both genders and different age ranges, from 10 primary health care units belonging to the ARS Centro [Regional Health Administration], from rural and urban areas.

Patients were selected semi-randomly as the first and last in consultation each day for 10 consecutive days of consultations (in order to avoid the bias of always having the same type of people), and on alternate days the physician consulted with or without the use of a white coat.

Exclusion criteria were considered as follows: under 18 years of age (in which case the questionnaire could be answered by the person accompanying him/her), illiterate patients and also patients whose general condition did not allow them to respond to the presented questionnaire. In the cases mentioned above, or in case of refusal, the physician could pass the questionnaire to the next patient (in case it was the first of the day) or to the first of the following day (if it was the last day), keeping the conditions aforementioned.

2.3 - Data collection instrument

The questionnaire addressed to the patient contained 2 scales duly translated and validated for the Portuguese language, whose authors gave the proper authorization for use in this study.

Each patient was asked about their age, gender, regular medication, literacy, level of education and professional activity. In the second part, they were asked about their satisfaction with the consultation and the medical knowledge perceived during the consultation, using a 0 to 4-point Likert scale. The "Trust in physician" scale - Portuguese version5, was applied, in which 11 items were presented, again using a 0 to 4-point Likert scale. This allows us to evaluate confidence in 3 aspects: the total trust of the physician, to which the 11 items correspond, trust in the relationship with the physician, to which only 6 items correspond (1, 4, 5, 7, 10 and 11) and finally the trust in the competence of the physician corresponding to 5 items (2,3,6,8 and 9). The JSPPPE-VP6 scale was applied in order to evaluate medical empathy, through 5 items to rank from 1 to 7 on a Likert scale. Finally, the patient's opinion on medical clothing was evaluated through 3 phrases: "1. Normal clothes worn by the physician make the environment more relaxed relative to the white coat. ", "2. It would be easier to communicate with a physician dressed in normal clothes. "e" 3. The white coat is the only attire acceptable for a physician.", with a scale equal to the previous one.

Regarding the questionnaire addressed to the physician, it was based on 2 simple yes/no questions with regard to having worn the white coat on a regular basis and 2 items related to his/her satisfaction and comfort during the consultation on a 0 to 4-point Likert scale.

2.4 - Data collection

The data collection took place from November 2018 to February 2019, in a period of 10 consecutive days, chosen by the physician. The questionnaire was delivered by the physician at the end of the consultation, after the patient signed the Informed Consent and filled out the self-completion questionnaire with the physician´s help in case of doubts or difficulties.

2.5 - Procedures prior to data collection

The study was authorized by the head of each health unit and the Ethics committee of the ARS do Centro [Regional Health Administration]

2.6 - Variables

The outcomes under study in this research, defined in protocol and unchanged after the field study, were as follows: Patient satisfaction, Total trust perceived by the patient, Confidence in the physician-patient relationship, Confidence in the physician's competences and Empathy perceived by the patient (main outcomes) and Knowledge perceived by the patient, Physician satisfaction and Physician comfort (secondary outcomes).

2.7- Statistical analysis

After a descriptive analysis, the normal distribution of numerical variables was tested using the Kolmogorov-Smirnov test. As the distribution of most variables was not normal, the non-parametric Mann-Whitney U tests were used to compare the numerical variables between the groups. The X2 test was used to compare the nominal variables. The value of p <0.05 was defined as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* A sample of 286 patients, of both sexes, of different ages and from health centers in both urban and rural areas belonging to the ARS Center was studied.

Exclusion Criteria:

* Age less than 18 years (in these cases the questionnaire can be answered by your companion).
* Illiterate patients.
* Patients whose general condition did not allow them to correctly answer the questionnaire presented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction: rating | 30 minutes
  A question about patient's satisfaction with the consultation rating from 0 to 4.
Trust | 30 minutes
  The use of the "Trust in physician" scale to evaluate patient trust in the medical-patient's relationship and in their medical competences.
Empathy | 30 minutes
  Empathy in the medical-patient's relationship evaluated through the Jefferson scale.

SECONDARY OUTCOMES:
Doctor's knowledge | 30 minutes
  Medical knowledge perceived by the patient evaluated through a question.
Doctor's satisfaction: question | 30 minutes
  A question that evaluated the doctor's satisfaction with the consultation.
Doctor's comfort: question | 30 minutes
  A question that evaluated the doctor's comfort with the consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Leonor Carreira, Principal Investigator — University of Coimbra
Locations (1):
- ARS Centro, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marques Caetano Carreira L, Dinis S, Correia A, Pereira A, Belo R, Madanelo I, Brito D, Gomes R, Monteiro L, Correia G, Maia C, Marques T, Sousa R, Abreu D, Matias C, Constantino L, Rosendo I. Does the white coat influence satisfaction, trust and empathy in the doctor-patient relationship in the General and Family Medicine consultation? Interventional study. BMJ Open. 2021 Dec 22;11(12):e031887. doi: 10.1136/bmjopen-2019-031887. PMID 34937710